CLINICAL TRIAL: NCT01173900
Title: Delivery, Uptake and Acceptability of HPV Vaccination in Tanzanian Girls
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Institute for Medical Research, Tanzania (Other Government); Ocean Road Cancer Institute, Tanzania (Unknown); Institut Català d' Oncologia, Spain (Unknown); Medical Research Council Social & Public Health Sciences Unit, UK (Unknown); International Union Against Cancer, Switzerland (Unknown)
Responsible Party: Principal Investigator, Deborah Watson-Jones, Dr, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MITU-001
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2011-11

CONDITIONS: Cervical Cancer
Keywords: human papillomavirus; vaccine; school girls; Tanzania; acceptability; vaccine coverage; Cervical cancer prevention
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Class-based delivery (Other): All girls attending standard 6 in schools selected for class-based vaccine delivery
  Interventions: Biological: Gardasil® HPV vaccine
- Age-based delivery (Other): All girls born in 1998 attending schools selected for age-based delivery
  Interventions: Biological: Gardasil® HPV vaccine

INTERVENTIONS:
Biological: Gardasil® HPV vaccine — 0.5 ml given at 0, 2, 6 months

SUMMARY:
The aims of this study are:

1. To determine feasibility of a school-based human papillomavirus (HPV) vaccination programme in Tanzania.
2. To measure the uptake and acceptability of two different vaccination strategies in rural and urban schools.
3. To examine the characteristics of accepters/refusers of vaccination and to identify reasons for acceptance, refusal or non-completion.
4. To measure the cost of implementing a school-based HPV vaccination programme in Tanzania.

DETAILED DESCRIPTION:
Vaccines against human papillomavirus infection, the primary cause of cervical cancer, are an attractive cervical cancer prevention strategy for resource poor settings which lack the infrastructure for establishing and maintaining complex screening programmes.Feasibility and costs of setting up and sustaining an HPV vaccination programme will depend on whether it can be added onto an existing health programme within schools, if one exists, or whether it has to be established as a separate health intervention. Other factors will also affect vaccine coverage. For example, uptake and overall effectiveness will be critically dependent on parental and community acceptability of a vaccine that prevents a sexually transmitted infection and how the vaccine is promoted and delivered by health-care providers will influence its uptake and acceptability.

This study will determine feasibility, uptake and acceptability of different delivery strategies of school-based HPV vaccination in Tanzania, examine factors related to acceptance or refusal of vaccination and measure the cost of implementing a school-based HPV vaccination programme in Tanzania.

Three doses of quadrivalent human papillomavirus (HPV) vaccine, (Gardasil®; Merck & Co) given at 0, 2 and 6 months, will be provided to 5000 primary school girls at 134 randomly selected schools in Mwanza Region in Tanzania. Selected schools will be randomly assigned to one of two delivery strategies (age-based or class-based) and coverage and acceptability of these vaccine delivery strategies will be compared. Qualitative research will be conducted before, during and after vaccination to examine barriers to vaccination and reasons for failure to complete vaccination as well as general community perceptions. To determine factors associated with refusal a case control study will be conducted on a 1:1 sample of 350 vaccine refusers and 350 accepters. The costs of introducing and scaling up HPV vaccines in schools will be estimated using established costing methods.

ELIGIBILITY:
Inclusion Criteria:

* female pupil
* attends selected school
* born in 1998 if enrolled in school selected for age-based delivery
* attending standard (class) 6 if enrolled in school selected for class-based delivery

Exclusion Criteria:

* has not previously received HPV vaccine
* has not participated in previous HPV vaccine trials

Min Age: 9 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5532 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Vaccine coverage by delivery strategy | Month 12
  Vaccine coverage will be estimated for each dose given and for those completing the full course of vaccination and compared by delivery strategy.
Vaccine coverage (dose 2) by delivery strategy | Month 5
Vaccine coverage (dose 1) by delivery strategy | Month 3

SECONDARY OUTCOMES:
Factors associated with refusal to vaccinate or to complete vaccination course | Month 12
  A case control study to determine factors associated with refusal will be conducted on a 1:1 sample of 350 vaccine refusers and 350 accepters.
Identification of barriers to HPV vaccination | Month 14
  Qualitative research will be conducted to examine barriers to vaccination and reasons for failure to complete vaccination.
Estimation of the costs of introducing and scaling up HPV vaccines in schools | Month 10
  Full financial and economic costs from the provider's perspective will be collected for the intervention. Total costs of a district vaccination programme and cost per urban school and rural school reached (if urban/rural differences are identified) and cost per fully-vaccinated girl will be estimated for the two alternative delivery strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah :L Watson-Jones, MD, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine; Richard J Hayes, DSC, Principal Investigator — London School of Hygiene and Tropical Medicine; John Changalucha, BSc, Principal Investigator — National Institute for Medical Research
Locations (1):
- National Institute for Medical Research, Mwanza, Tanzania

REFERENCES:
- [Derived] Quentin W, Terris-Prestholt F, Changalucha J, Soteli S, Edmunds WJ, Hutubessy R, Ross DA, Kapiga S, Hayes R, Watson-Jones D. Costs of delivering human papillomavirus vaccination to schoolgirls in Mwanza Region, Tanzania. BMC Med. 2012 Nov 13;10:137. doi: 10.1186/1741-7015-10-137. PMID 23148516
- [Derived] Watson-Jones D, Baisley K, Ponsiano R, Lemme F, Remes P, Ross D, Kapiga S, Mayaud P, de Sanjose S, Wight D, Changalucha J, Hayes R. Human papillomavirus vaccination in Tanzanian schoolgirls: cluster-randomized trial comparing 2 vaccine-delivery strategies. J Infect Dis. 2012 Sep 1;206(5):678-86. doi: 10.1093/infdis/jis407. Epub 2012 Jun 18. PMID 22711908